CLINICAL TRIAL: NCT04264507
Title: Prevalence and Outcomes of Acute Kidney Injury Among Medical ICU Patients in Assiut University Hospitals
Brief Title: Prevalence , Risk Factors and Outcomes of AKI in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, manal adel ahmed, resident doctor, Assiut University
Other Study IDs: Epidemiology of aki in icu
Record Dates: First submitted 2020-01-16; First posted 2020-02-11 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early recognition of AKI is essential to ensure prompt and appropriate management, and to avoid progression to late stages of the disease (2) AKI requiring renal replacement therapy occurs in 5-6% of ICU patients, with an extremely high in hospital mortality rate of 60%.6 It is estimated that about 2 million people die of AKI every year. Those who survive AKI have a higher risk for later development of CKD(3). Epidemiology of AKI is understudied in developing countries so further studies are needed to estimate the burden of AKI among ICU patients.

Few studies about the epidemiology of AKI in Egypt were done;

DETAILED DESCRIPTION:
Acute kidney injury is a sudden episode of kidney failure or damage that happens within a few hours or days. According to KDIGO (kidney disease improving global outcomes) criteria: AKI is defined as any of the following: Increase in serum creatinine by 0.3mg/dL or more within 48 hours or. Increase in serum creatinine to 1.5 times baseline or more within the last 7 days or. Urine output less than 0.5 mL/kg/h for 6 hours(1). Kidney Injury (AKI) affects over 13 million people per year globally and results in 1.7 million deaths. Recent hospital studies in the developed world report AKI in 3.2-9.6% of admissions, with overall in-hospital mortality around 20%, and up to 50% in ICU patients.

Early recognition of AKI is essential to ensure prompt and appropriate management, and to avoid progression to late stages of the disease (2) AKI requiring renal replacement therapy occurs in 5-6% of ICU patients, with an extremely high in hospital mortality rate of 60%.6 It is estimated that about 2 million people die of AKI every year. Those who survive AKI have a higher risk for later development of CKD(3). Epidemiology of AKI is understudied in developing countries so further studies are needed to estimate the burden of AKI among ICU patients.

Few studies about the epidemiology of AKI in Egypt were done; Samar Abd ElHafeez e,tal 2017 found in a multicenter study of over 500 consecutive patients admitted to ICUs in Alexandria Teaching Hospitals in Egypt, that about 40% of patients admitted to ICU had AKI at presentation, and a similar proportion of those who were AKI-free on admission developed AKI during their ICU stay (4) .

Up to our knowledge, there are no sufficient data about the epidemiology of AKI in upper Egypt

ELIGIBILITY:
Inclusion Criteria:

* All patients >18 years admitted to medical ICU in Internal Medicine Department with critical medical conditions who develop AKI during hospital admission or presented with AKI

Exclusion Criteria:

* Patients with ESRD on regular dialysis ,Patients with stage 4 or 5 non-dialysis if the condition proven to be progression of the already known diagnosis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: cases of AKI admitted to ICU in internal medicine department or developed AKI during hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of AKI patients admitted to medical ICU in assiut university hospitals | One year
  Number of patients addimmted or developed aki during stay in icu

SECONDARY OUTCOMES:
The proportion of risk factor of AKI | one year
  Most common risk factors for aki in ice patients

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Hosny, Doctor, Study Director — Assiut University
Locations (1):
- Assiut university Hospital, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Summary of Recommendation Statements. Kidney Int Suppl (2011). 2012 Mar;2(1):8-12. doi: 10.1038/kisup.2012.7. No abstract available. PMID 25018916
- See also: Summary of Recommendation Statements. Kidney Int Suppl — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4089654/